CLINICAL TRIAL: NCT02402348
Title: Pilot Study of Metformin (MF) IN HNSCC (Head and Neck Squamous Cell Carcinoma) as Window Trial Design in Operable HNSCC, to Investigate the Effects of MF, Tumor Genotype and MF Genotype Interactions, on Tumor Metabolism and Anoikis
Brief Title: Pilot Study of Metformin in HNSCC to Investigate the Effects of MF, Tumor Genotype and MF-genotype Interactions, on Tumor Metabolism and Anoikis
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding not available, PI left institution
Sponsor: West Virginia University (Other)
Collaborators: West Virginia Clinical and Translational Science Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WV011614
Record Dates: First submitted 2015-03-24; First posted 2015-03-30 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Cancer of Head and Neck
Keywords: head and neck squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): Metformin 850 mg orally once a day for 3 days, then 850 mg orally twice daily starting day 4 until 24hrs before surgery.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin
  Other Names: Glucophage

SUMMARY:
The study researchers want to look at the overall effects that Metformin may have on the tumor characteristics of Head and Neck cancer cells as well as the interactions that Metformin has on the growth or death of tumor cells.

DETAILED DESCRIPTION:
Subjects will sign informed consent and have their medical records reviewed, a physical exam and blood taken for lab tests and a biopsy of the cancer will be taken to determine eligibility for the study.

Following enrollment, the subject will begin to take Metformin at a dosage of 850 mg daily on Days 1 through 3 (in the mornings with breakfast). On day 3 the study team will call to see if the subject is tolerating the Metformin.

If tolerated, then the dose will increase to 850 mg twice a day (with breakfast and dinner) on starting on Day 4.

This dose is to continue until 24 hours prior to surgery, with a minimum of 14 days but can be extended until 28 days dependent on planned surgery date.

The study team will provide the subject with the Metformin and a study diary to record when they take their pills and if there are any issues to communicate to the physician. They will also be contacted by phone or planned visit days to see how their body is tolerating the Metformin throughout their treatment (approximately every 3 days).

On Day 14 plus or minus 3 days (or 2 weeks after staring Metformin) and immediately prior to surgery, the physician will collect a blood sample.

On the day of surgery, the surgeon will remove the tumor and send it to the lab for evaluation as part of standard cancer care. They will also collect an additional biopsy of the tumor for research purposes to test the effects of Metformin on the tumor cells.

The subjects will be followed for 30 days after their surgery.

The blood and tumor samples collected will be sent to a research lab at WVU for to test the effect of Metformin, tumor genotype and Metformin genotype interactions on critical tumor cell metabolic parameters and also on anoikis-sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed HNSCC Stage II-IVB (T1N1-3, T2-3, N0-3, M0) OR Patients with suspected Stage II-IVB tumor as determined by clinical examination or noted via imaging.
* Planned complete resection of the primary tumor.
* Age >= 18 years.
* ECOG performance status of 0 or 1
* Adequate hepatic, renal, and bone marrow function

Exclusion Criteria:

* Prior therapy for head and neck cancer
* Candidates for neo-adjuvant chemotherapy or chemo-radiation therapy for curative intent.
* Co-existing malignancy or malignancies diagnosed within the last 3 years with the exception of basal cell carcinoma or in situ cervical cancer.
* History of diabetes mellitus or taking any medications indicated for diabetes mellitus treatment
* Contraindication to metformin including hypersensitivity or allergic reaction
* Active diagnosis of Alcoholism
* Congestive heart failure requiring pharmacologic treatment.
* BMI < 25
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Tumor cell death estimated by percentage | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Fancy, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Hospitals - Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frisch SM, Schaller M, Cieply B. Mechanisms that link the oncogenic epithelial-mesenchymal transition to suppression of anoikis. J Cell Sci. 2013 Jan 1;126(Pt 1):21-9. doi: 10.1242/jcs.120907. PMID 23516327
- [Background] Sandulache VC, Hamblin JS, Skinner HD, Kubik MW, Myers JN, Zevallos JP. Association between metformin use and improved survival in patients with laryngeal squamous cell carcinoma. Head Neck. 2014 Jul;36(7):1039-43. doi: 10.1002/hed.23409. Epub 2014 Jan 29. PMID 23784886
- [Background] Bonanni B, Puntoni M, Cazzaniga M, Pruneri G, Serrano D, Guerrieri-Gonzaga A, Gennari A, Trabacca MS, Galimberti V, Veronesi P, Johansson H, Aristarco V, Bassi F, Luini A, Lazzeroni M, Varricchio C, Viale G, Bruzzi P, Decensi A. Dual effect of metformin on breast cancer proliferation in a randomized presurgical trial. J Clin Oncol. 2012 Jul 20;30(21):2593-600. doi: 10.1200/JCO.2011.39.3769. Epub 2012 May 7. PMID 22564993